CLINICAL TRIAL: NCT02579499
Title: Low-Density Lipoprotein Cholesterol-targeting Statin Therapy Versus the Intensity-based Statin Therapy in Patients With Coronary Artery Disease: a Randomized Comparison Trial
Brief Title: Low-Density Lipoprotein Cholesterol-targeting Statin Therapy Versus the Intensity-based Statin Therapy in Patients With Coronary Artery Disease
Acronym: LODESTAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0713
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Diseasse
Keywords: Coronary artery disease; LDL choelsterol; Statin
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixed high-potent statin group (Active Comparator): According to 2013 ACC/AHA guideline, patients will be received high-intensity statin therapy (atorvastatin 40mg or rosuvastatin 20mg) regardless of their baseline LDL-C levels.
  Interventions: Drug: fixed high potent statin therapy
- Targeted LDL-C goal statin group (Experimental): Patients will be tiltrated statin intensity guided by follow-up LDL-C level
  Interventions: Drug: targeted LDL-C goal statin

INTERVENTIONS:
Drug: fixed high potent statin therapy — Patients assigned fixed high-potent statin group will be received high-intensity statin therapy (atorvastatin 40mg or rosuvastatin 20mg) regardless of their baseline LDL-C levels, and maintain high-intensity statin therapy regardless of their follow-up LDL-C level.
  Arms: Fixed high-potent statin group
Drug: targeted LDL-C goal statin — 1. Statin naïve patients: Patients will be received moderate intensity statin therapy (atorvastatin 20mg or rosuvastatin 10mg)
  2. Patients already received statin therapy
     * Baseline LDL-C <70mg: same intensity of statin therapy
     * Baseline LDL-C≥70mg: uptiltrated statin therapy Patients will be tiltrated statin intensity guided by follow-up LDL-C level ( Attained LDL-C < 50mg/dL : down regulated intensity statin therapy, 50mg/dL ≤ Attained LDL-C < 70g/dL: maintain current intensity statin therapy, Attained LDL-C ≥ 70mg/dL: up regulated intensity statin therapy)
  Arms: Targeted LDL-C goal statin group

SUMMARY:
To compare clinical safety & efficacy of fixed-high potent statin therapy (according to 2013 ACC/AHA guideline) vs. targeted LDL-C goal statin therapy (LDL<70mg/dL) for secondary prevention. Total 4400 patients with coronary artery disease patients requiring statin treatment were categorized fixed high-potent statin group and targeted LDL-C group. The investigators will compare primary endpoint (major adverse cardiac and cerebrovascular event (MACCE)) and secondary endpoint (1. New onset diabetes mellitus after randomization, 2. Hospitalization due to heart failure, 3. Deep vein thrombosis or Pulmonary thromboembolism, 4. Percutaneous trans-luminal angioplasty on peripheral artery obstructive disease, 5. Aortic intervention or operation, 6. ESRD with renal replacement therapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients clinically diagnosed with coronary artery disease including stable angina, unstable angina, acute non-ST elevation myocardial infarction and acute ST elevation myocardial infarction
* Patients with signed informed consent

Exclusion Criteria:

* Pregnant women or women with potential childbearing
* Patients severe adverse events or hypersensitive to statin or patients with multi-drug allergy.
* Who had received drug that have a drug interaction with statin (strong inhibitor of cytochrome p-450 3A4 or 2C9)
* Patients with risk factors for myopathy with hereditary muscle disorder, hypothyroidism, alcohol use disorder, severe hepatic dysfunction (3 times normal reference values) or rhabdomyolysis
* Life expectancy < 3 years
* Patient with who can not be followed up for more than 1 year
* Patients who cannot understand or read the consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4400 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 3 years

SECONDARY OUTCOMES:
numer of other adverse clinical events | 3 years
  1. New onset diabetes mellitus after randomization
  2. Hospitalization due to heart failure
  3. Deep vein thrombosis or Pulmonary thromboembolism
  4. Percutaneous trans-luminal angioplasty on peripheral artery obstructive disease
  5. Aortic intervention or operation
  6. ESRD with renal replacement therapy
  7. Discontinuation of study drugs due to intolerance
  8. Cataract operation
  9. Composite of laboratory abnormality (ALT >3x ULN, CK >5x ULN, or elevation in creatinine)

CONTACTS AND LOCATIONS:
Overall Officials: MYEONG-KI HONG, MD, PhD, Principal Investigator — Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Hong SJ, Lee YJ, Kang WC, Hong BK, Lee JY, Lee JB, Yang TH, Yoon J, Lee SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK; LODESTAR investigators. Effect of rosuvastatin versus atorvastatin on new-onset diabetes mellitus in patients treated with high-intensity statin therapy for coronary artery disease: a post-hoc analysis from the LODESTAR randomized clinical trial. Cardiovasc Diabetol. 2024 Aug 7;23(1):287. doi: 10.1186/s12933-024-02386-w. PMID 39113067
- [Derived] Lee SJ, Lee JB, Yang TH, Kang WC, Lee JY, Lee YJ, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Hong BK, Choi D, Yoon J, Jang Y, Hong MK; LODESTAR investigators. Treat-to-target or high-intensity statin treatment in older adults with coronary artery disease: a post hoc analysis of the LODESTAR trial. Age Ageing. 2024 Jul 2;53(7):afae132. doi: 10.1093/ageing/afae132. PMID 38965031
- [Derived] Lee YJ, Hong SJ, Kang WC, Hong BK, Lee JY, Lee JB, Cho HJ, Yoon J, Lee SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK; LODESTAR investigators. Rosuvastatin versus atorvastatin treatment in adults with coronary artery disease: secondary analysis of the randomised LODESTAR trial. BMJ. 2023 Oct 18;383:e075837. doi: 10.1136/bmj-2023-075837. PMID 37852649
- [Derived] Lee SJ, Kang WC, Lee JY, Lee JB, Yang TH, Yoon J, Lee YJ, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Hong BK, Jang Y, Hong MK; LODESTAR Investigators. Treat-to-target versus high-intensity statin treatment in patients with or without diabetes mellitus: a pre-specified analysis from the LODESTAR trial. EClinicalMedicine. 2023 Sep 20;64:102227. doi: 10.1016/j.eclinm.2023.102227. eCollection 2023 Oct. PMID 37767195
- [Derived] Hong SJ, Lee YJ, Lee SJ, Hong BK, Kang WC, Lee JY, Lee JB, Yang TH, Yoon J, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK; LODESTAR Investigators. Treat-to-Target or High-Intensity Statin in Patients With Coronary Artery Disease: A Randomized Clinical Trial. JAMA. 2023 Apr 4;329(13):1078-1087. doi: 10.1001/jama.2023.2487. PMID 36877807